CLINICAL TRIAL: NCT04243603
Title: Treatment Effects of Internet-based Emotion Regulation Individual Therapy for Adolescents (ERITA) Added to Treatment as Usual in Young People With Non-Suicidal Self-Injury - (TEENS) Feasibility Trial
Brief Title: Effects of Internet-based ERITA Added to TAU in Young People With Non-Suicidal Self-Injury (TEENS) Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Britt Reuter Morthorst, Principal investigator, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19042904
Record Dates: First submitted 2020-01-16; First posted 2020-01-28 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Non-suicidal Self-injury
Keywords: Non-suicidal Self-injury; Internet-based intervention
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Single-center, feasibility trial including a randomization procedure in a parallel group design with blinded outcome assessment.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, a blinding of participants and therapists (intervention providers) is not possible. Blinded outcome assessment and data management will be performed. Statistical analyses will be performed by two blinded statisticians presenting independent reports. Based on the two blinded conclusions, two abstracts will be written and published (on a website).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based ERITA-DK (Experimental): ERITA is a youth-adapted version of Emotion Regulation Group Therapy (ERGT), based on cognitive behavioral therapy (CBT), dialectical behavior therapy (DBT), and Acceptance and Commitment Therapy (ACT), which encounters emotional recognition and regulation, crisis strategies and skills training. The ERITA intervention is provided as add-on to TAU and consists of 12 weeks, manualized, therapist guided internet-based therapy. The intervention also provides six modules for the parents focusing on NSSI and other risk-taking behaviors, emotional awareness, and validation skills. The participants must complete one module every week while the parents must complete a module every second week. A mobile app is available to complement the online treatment. The app includes reminders of homework and skills and allows to report on both self-destructive behaviors and impulses daily.
  Interventions: Behavioral: Internet-based Emotion Regulation Individual Therapy for Adolescents (ERITA-DK)
- Treatment as Usual (TAU) (Active Comparator): Child and Adolescent Mental Health Services (CAMHS) offer specialized treatment for children and adolescents. TAU encounters a variety of clinical treatment and assessment offers, representing a highly inhomogeneous group of treatments, for instance: Pharmacological treatment, Family-Based Treatment (FBT), Cognitive Behavioral Therapy, supportive counselling and psychoeducation. Throughout the trial course the treatment responsibility is handled by clinicians providing TAU.
  Interventions: Behavioral: Internet-based Emotion Regulation Individual Therapy for Adolescents (ERITA-DK)

INTERVENTIONS:
Behavioral: Internet-based Emotion Regulation Individual Therapy for Adolescents (ERITA-DK) — Please see description of experimental arm (arm one)

SUMMARY:
There has been a significant increase in non-suicidal self-injury the last decades especially among young people and treatment initiative are sparse. We aim to assess the feasibility of methods, procedures, and safety of internet-based Emotion Regulation Individual Therapy for Adolescents (ERITA) as add on to treatment as usual (TAU) in 13-17-year-old patients with non-suicidal self-injury referred to psychiatric services.

DETAILED DESCRIPTION:
Non-suicidal self-injury has disseminated almost epidemically through the last decades in young persons. There is no evidence of any experimental treatment for non-suicidal self-injury in adolescents, superior to treatment as usual. Patients with stigmatizing illness such as non-suicidal self-injury may find internet-based interventions more acceptable. The study is a feasibility trial, with a randomization procedure in a parallel group design. Patients will be recruited from Child- and Adolescent Mental Health Services (age 13 to 17 years). The experimental intervention is internet-based, and therapist guided; ERITA consists of online Emotion Regulation Individual Therapy for Adolescents (ERITA) as add-on to treatment as usual. Treatment as usual is provided by multidisciplinary teams in nine outpatient clinics within Child and Adolescent Mental Health Services in the Capital Region of Denmark. Feasibility of recruitment and trial procedures will be monitored as well as explorative clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 5 non-suicidal self-injury episodes in the past year and ≥ 1 non-suicidal self-injury episodes in the past month (DSM-5 criteria for a diagnosis of non-suicidal self-injury disorder in terms of frequency of NSSI).
* Age-appropriate literacy.
* Having at least one parent committing to participate in the parent program.
* Informed consent from parents/legal caretakers.

Exclusion Criteria:

* Imminent suicidal risk assessed by clinicians during routine screening procedure (rated as no risk, elevated risk, imminent risk) in need of admission or other life saving strategies.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-01-22 (Actual)

PRIMARY OUTCOMES:
Completion of follow-up | End of treatment at 12 weeks
  Completion of follow-up will be defined as completing at least one clinical outcome (non-suicidal self-injury events) at end of intervention. If the number participants with completed outcomes is 26 out of 30, the fraction will be 87%, 95% CI 75% to 99%. A follow-up fraction of 87% or more will be acceptable for a future trial while a fraction below 75% will impose serious problems of interpreting the trial result in a future large pragmatic trial.
The fraction of eligible participants who consent to inclusion and randomization | End of treatment at 12 weeks
  We will determine the fraction of potential participants as the number of eligible persons compared to the number of randomized persons. If the number of participants randomized out of the number of eligible persons is 30 out of 75, the fraction will be 40%, 95% confidence interval (CI) will be: 29% to 51%. A randomization fraction of 29% or more will be acceptable for a future trial, while a fraction below 29% will impose serious problems of recruitment for a future large pragmatic trial.
Compliance | End of treatment at 12 weeks
  Compliance with the experimental intervention will be defined as completing at least six of 12 ERITA sessions. ERITA will automatically register time for login and save the exercises that have been completed. If the number of compliant experimental participants is 11 out of 15, the fraction will be 73%, 95% CI 51% to 96%. A compliance fraction of 51% or more will be acceptable for a future trial while a fraction below 51% will impose serious problems of interpreting the trial result in a future large pragmatic trial.
Non-suicidal self-injury as explorative primary clinical outcome | End of treatment at 12 weeks
  Non-suicidal self-injury, assessed at baseline and end of therapy (12 weeks) by blinded outcome assessment by phone with Deliberate Self-Harm Inventory (DSHI-Y)

SECONDARY OUTCOMES:
Quality of life as explorative secondary clinical outcomes | End of treatment at 12 weeks
  Quality of life at 12 weeks, assessed with Kidscreen-10. 5-point Likert scale, range: not at all, a little, modearte, much, very much.
Symptoms of depression, anxiety and stress as explorative secondary clinical outcomes | End of treatment at 12 weeks
  Symptoms of depression, anxiety and stress at 12 weeks, assessed with Depression Anxiety Stress Scale (DASS-21). 4-point Likert scale, range: did not apply to me, applied to me to some degree, applied to me to a considerable degree, applied to me much/most of the time. Totale range for subscores: 0-42. Higher scores reflects worse outcome.
Non-suicidal self-injury as dichotomous variables as explorative secondary clinical outcome | End of treatment at 12 weeks
  Non-suicidal self-injury as dichotomous variables (Yes/No)
Number of sick days the last month as explorative secondary clinical outcome | End of treatment at 12 weeks
  Number of sick days the last month

OTHER OUTCOMES:
Difficulties in emotion regulation as further explorative clinical outcome | At end of treatment and once a week for 12 weeks
  Difficulties in emotion regulation, assessed weekly during 12 weeks with Difficulties in Emotion Regulation Scale (DERS-16). 5-point Likert scale, range: almost never, some times, half of the time, most of the time, all the time. Total scores range from 16 to 80, with higher scores reflecting grater levels of emotion dysregulation.
Indirect self-destructive behaviours as further explorative clinical outcome | End of treatment at 12 weeks
  Indirect self-destructive behaviours at 12 weeks, assessed with Borderline Symptom List (BSL-supplement). 5-point Likert scale, range: not at all, once, 2-3 times, 4-6 times, daily or more often. Total scores range from 0-44 and higher scores reflect worse outcome.
Suicidal ideations, plans and actions as further explorative clinical outcome | End of treatment at 12 weeks
  Suicidal ideations, plans and actions at 12 weeks, assessed with Columbia (C-SSRS). Dichotomous outcome yes/no; if yes intensity is rated on a 5-point Likert scale, total score range: 2-25. Higher scores reflect worse outcome.
Parents' ability to cope with children's negative emotions as further explorative clinical outcome | After week six and week 12
  Adolescent's perception of Parents' ability to cope with children's negative emotions at 6 weeks and 12 weeks, assessed with The Coping with Children's Negative Emotions Scale (CCNES-APP). 7-point Likert scale, Range from very unlikely to very likely. Six Sub scales with total score range: 0-42. The sub scale are inversely related.
Parents' perceived ability to cope with children's negative emotions as further explorative clinical outcome | After week six and week 12
  Parents' perceived ability to cope with children's negative emotions at 6 weeks and 12 weeks, assessed with The Coping with Children's Negative Emotions Scale Adolescent (CCNES-A). 7-point Likert scale, Range from very unlikely to very likely. Six Sub scales with total score range: 0-42. The sub scale are inversely related.
Adverse Events as further explorative clinical outcome | After week 4, 8, and 12
  Adverse Events 4, 8 and 12 weeks assessed with Negative Effects Questionnaire (NEQ). Dichotomous outcomes as yes/no; if yes then a 5-point Likert scale of the impact, range not at all, a little, moderately, much, very much. The total score range 0-80. Higher scores reflect worse outcome.
Strengths and difficulties as further explorative clinical outcome | After week 4, 8, and 12
  Strengths and difficulties assessed by Strengths and difficulties questionnaire (SDQ) at 4, 8, and 12 weeks. 3-point Likert scale, range: doesn't fit, fits moderately, fits very much. Total score range 0-40. Sub scales of strengths and difficulties that are inversely related.
Working alliance with online therapist as further explorative clinical outcome | After week 4, 8, and 12
  Working alliance with online therapist assessed with Working Alliance Inventory (WAI-SR). 5-point Likert scale, range: seldom, some times, fairly often, very often, always. Total score range 12-60. Higher scores reflect higher working alliance/better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Katrine Pagsberg, Professor, Study Director — Child & Adolescent Mental Health Services Capital Region of Denmark
Locations (1):
- Team for Self-injury, Child and Adolescent Mental Health Services, B195, Copenhagen, Ø, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsen MH, Morthorst B, Pagsberg AK, Heinrichsen M, Mohl B, Rubaek L, Bjureberg J, Simonsson O, Lindschou J, Gluud C, Jakobsen JC. An Internet-based emotion regulation intervention versus no intervention for non-suicidal self-injury in adolescents: a statistical analysis plan for a feasibility randomised clinical trial. Trials. 2021 Jul 16;22(1):456. doi: 10.1186/s13063-021-05406-2. PMID 34271984
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Interventions for self-harm in children and adolescents. Cochrane Database Syst Rev. 2021 Mar 7;3(3):CD013667. doi: 10.1002/14651858.CD013667.pub2. PMID 33677832
- [Derived] Morthorst B, Rubaek L, Lindschou J, Jakobsen JC, Gluud C, Bjureberg J, Hellner C, Mohl B, Pagsberg AK. An internet-based emotion regulation intervention versus no intervention for nonsuicidal self-injury in adolescents: study protocol for a feasibility trial. Pilot Feasibility Stud. 2021 Feb 6;7(1):44. doi: 10.1186/s40814-021-00785-4. PMID 33549128